CLINICAL TRIAL: NCT05258045
Title: Is Mediastinal Blood Pool SUV Ratio Valid in Identification of Malignancy in Comparison to Liver SUV Ratio?
Brief Title: Validity of Mediastinal Blood Pool SUV Ratio
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zainab Fathy Mohammed, Resident doctor, Assiut University
Other Study IDs: PET/CT in malignancy
Record Dates: First submitted 2022-02-22; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Validity of Blood Pool SUV Ratio in Identification of Malignancy in Case of Diseased Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- SUV ratio of mediastinal blood pool to the lesion and SUV ratio of liver to lesion: Avidity of SUV of blood pool
  Interventions: Radiation: F18 FDG

INTERVENTIONS:
Radiation: F18 FDG — Radioactive material

SUMMARY:
-Validity of blood pool SUV ratio in identification of malignancy in case of diseased liver.

DETAILED DESCRIPTION:
PET/CT is the functional imaging tool that can measure increased glucose metabolism in cancer tissues by using flourine 18 FDG which is FDA approved and used routinely in identification of malignant lesions , staging and restaging of many malignancy like lymphoma, breast cancer, lung cancer and cancer colon.

In clinical routine, SUV is often used to determine the glucose metabolism in tumours by 18F-FDG PET/CT. And can be further normalised to SUVs in reference regions resulting in a SUV ratio (SUV ratio).in routine work SUV of the lesion is normalised to SUV of the liver , but this not used if the liver is diseased like as liver cirrhosis or liver metastases , so SUV ratio of lesion to mediastinal blood pool and SUV ratio of the lesion to liver will be measured in correlation to pathology to assess validity of SUV of mediastinal blood pool.

ELIGIBILITY:
Inclusion Criteria:

* This study will include cancer pt who did PET/CT scan who presented to nuclear medicine unit during the period from 2021 until the end of the study.

Exclusion Criteria:

* Severely ill patient
* Pt with glucose level above 200

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Cross sectional study prospective and retrospective
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
-Validity of blood pool suv ratio in identification of malignancy in case of diseased liver. | One year
  PET/CT is the functional imaging tool that can measure increased glucose metabolism in cancer tissues by using flourine 18 FDG which is FDA approved and used routinely in identification of malignant lesions , staging and restaging of many maligancy like lymphoma, breast cancer, lung cancer and cancer colon.
  In clinical routine, SUV is often used to determine the glucose metabolism in tumours by 18F-FDG PET/CT. And can be further normalised to SUVs in reference regions resulting in a SUV ratio (SUV ratio).in routine work SUV of the lesion is normalised to SUV of the liver , but this not used if the liver is diseased like as liver cirrhosis or liver metastases , so SUV ratio of lesion to mediastinal blood pool and SUV ratio of the lesion to liver will be measured in correlation to pathology to assess validity of SUV of mediastinal blood pool.